CLINICAL TRIAL: NCT06971458
Title: Endometrioma Ethanol Sclerotherapy and Its Effect on Ovarian Function and Fertility Treatment Outcome - Prospective Cohort Study Protocol
Brief Title: Endometrioma Ethanol Sclerotherapy - Prospective Cohort Study Protocol
Status: Recruiting | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0008-22-HYMC
Record Dates: First submitted 2023-03-07; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: IVF; Endometrioma
MeSH Terms: conditions — Endometriosis | interventions — Sclerotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- women with endometrioma size of 25-100 mm: Prospective cohort study including women with endometrioma size of 25-100 mm who will undergo ultrasound (US)-guided sclerotherapy. IVF treatment can be done about a month afterwards.
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Sclerotherapy — ultrasound (US)-guided sclerotherapy for the treatment of ovarian endometrioma

SUMMARY:
Ovarian endometriomas are cystic masses lined with endometrial tissue that contains fluid arising from a collection of menstrual debris. Ovarian endometriomas clinical manifestations includes pelvic pain, dysmenorrhea, dysfunctional uterine bleeding, and infertility.

Endometriomas are most commonly treated either medically or by surgical excision.

Ultrasonography (US)-guided aspiration and sclerotherapy is a new approach. Its mechanism of action is believed to be destruction of the inner epithelial lining, which is followed by inflammation and fibrosis, eventually resulting in regression of the cyst. The main advantage in this approach is the avoidance of collateral damage to the ovary.

DETAILED DESCRIPTION:
Endometriosis is a disease of the female reproductive system in which cells similar to those in the endometrium grow outside the uterus. Endometriosis prevalence is estimated to be around 10%, and even higher among women with infertility.

Endometriosis can involve any pelvic organ and in rare cases it may also occur in other parts of the body.

Ovarian endometriomas are cystic masses lined with endometrial tissue that contains fluid arising from a collection of menstrual debris. Ovarian endometriomas clinical manifestations includes pelvic pain, dysmenorrhea, dysfunctional uterine bleeding, and infertility.

Endometriomas are most commonly treated either medically or by surgical excision. Surgical excision is considered the standard therapy when pain is not controlled well by medication or when malignancy is being suspected. However, deterioration in the ovarian reserve after cystectomy is inevitable due to the removal of normal ovarian tissue adjacent to the endometrioma, and the possibility of excessive electrocoagulation for hemostasis.

Ultrasonography (US)-guided aspiration and sclerotherapy is a new approach. Its mechanism of action is believed to be destruction of the inner epithelial lining, which is followed by inflammation and fibrosis, eventually resulting in regression of the cyst. The main advantage in this approach is the avoidance of collateral damage to the ovary. There are still no guidelines suggesting US-guided sclerotherapy for endometrioma, although it has been used worldwide over the years since its introduction, and is reported to be an effective therapeutic option for endometriosis-associated pain and infertility. There are several reports of a higher oocyte number and higher pregnancy rate in IVF treatments after sclerotherapy in comparison with IVF after cystectomy. There is also a report of higher pregnancy rate in IVF treatments after sclerotherapy in comparison with leaving the endometrioma in-situ.

The procedure is done in an ambulatory arrangement under general anesthesia. Antibiotic prophylaxis with cefazolin 2g is administrated before beginning of the procedure. First step is (US)-guided aspiration of the endometrioma content. A sample of the aspirated content is sent to cytology test. Second, the cyst is flushed with normal saline. Third, the cyst is filled with 95% ethanol. The ethanol is suspended for 10-15 minutes inside the cyst capsule and then aspirated

ELIGIBILITY:
Inclusion Criteria:

A woman with endometrioma with a diameter of 25-100 mm

Exclusion Criteria:

* Other causes of infertility (sperm disorder, ovulation disorder, uterine disorder, mechanical factor, poor ovarian reserve)

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females only
Study Population: A woman with endometrioma with a diameter of 25-100 mm who is intended for IVF treatment to achieve pregnancy or for medical preservation/by choice.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of | 3 Years
  ultrasound (US)-guided sclerotherapy for the treatment of ovarian endometrioma effect on ovarian function and fertility treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Einat Shalom-Paz, Prof, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel